CLINICAL TRIAL: NCT00758589
Title: A Double-blind, Randomised, Parallel Group, Multicentre Phase IIb, Placebo-Controlled, 1 Month Dose Response Study of AZD1981 in Asthma Patients Uncontrolled on Inhaled Steroids
Brief Title: One Month Dose Response Study of AZD1981 in Asthma Patients Uncontrolled on Inhaled Steroids
Acronym: OLIVE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D9830C00004
Record Dates: First submitted 2008-09-23; First posted 2008-09-25 (Estimated); Results first posted 2013-12-13 (Estimated); Last update posted 2014-02-26 (Estimated); Status verified 2014-01

CONDITIONS: Asthma
Keywords: Asthma
MeSH Terms: conditions — Asthma | interventions — AZD1981

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- AZD1981 50 mg (Experimental): AZD1981 50 mg Twice Daily (Bid)
  Interventions: Drug: AZD1981
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo
- AZD1981 400 mg (Experimental): AZD1981 400 mg Twice Daily (Bid)
  Interventions: Drug: AZD1981
- AZD1981 1000 mg (Experimental): AZD1981 1000 mg Twice Daily (Bid)
  Interventions: Drug: AZD1981

INTERVENTIONS:
Drug: AZD1981 — Oral tablet, 50 mg twice daily
  Arms: AZD1981 50 mg
Drug: AZD1981 — Oral tablet, 400 mg twice daily
  Arms: AZD1981 400 mg
Drug: AZD1981 — Oral tablet, 1000 mg twice daily
  Arms: AZD1981 1000 mg
Drug: Placebo
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate efficacy of AZD1981 in uncontrolled asthmatic patients on maintenance inhaled glucocorticosteroids.

ELIGIBILITY:
Inclusion Criteria:

* Six months history of asthma
* Daily use of inhaled glucocorticosteroids
* FEV1 40-85% of predicted normal
* Reversibility; increase in FEV1 more than 12% and 200 mL post-bronchodilator

Exclusion Criteria:

* Other clinically relevant disease or disorders
* History of smoking of more than 10 pack years
* Respiratory infection within 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 368 (Actual)
Dates: Start 2008-09; Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Kuna, Principal Investigator — University of Lodz, Lodz, Poland
Locations (21):
- Argentina (4):
  - Research Site, Buenos Aires, Argentina
  - Research Site, Quilmes, Buenos Aires
  - Research Site, Santa Fe, Santa Fe Province
  - Research Site, San Miguel de Tucumán, Tucumán Province
- Brazil (4):
  - Research Site, Porto Alegre, Brasil
  - Research Site, Rio de Janeiro, Rio de Janeiro
  - Research Site, Santo André, São Paulo
  - Research Site, São Paulo, São Paulo
- Costa Rica (2):
  - Research Site, Barrio Los Yoses, Provincia de San José
  - Research Site, San Francisco de Dos Ríos, Provincia de San José
- Poland (11):
  - Research Site, Bialystok
  - Research Site, Bydgoszcz
  - Research Site, Gdalsk
  - Research Site, Kielce
  - Research Site, Krakow
  - Research Site, Lublin
  - Research Site, Poznal
  - Research Site, Szczecin
  - Research Site, Tarnów
  - Research Site, Turek
  - Research Site, Wroclaw

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 510 patients enrolled, 368 were allocated to treatment and 350 completed the study. First patient entered the study on 16 September 2008 and the last patient finished the study on 13 July 2009.
Groups:
- AZD1981 50 mg Twice Daily (Bid): AZD1981 oral tablet 50 mg, twice daily
- AZD1981 400 mg Twice Daily (Bid): AZD1981 oral tablet 400 mg, twice daily
- AZD1981 1000 mg Twice Daily (Bid): AZD1981 oral tablet 1000 mg, twice daily
- Placebo: placebo oral tablet, twice daily
Period: Overall Study
Arm/Group | AZD1981 50 mg Twice Daily (Bid) | AZD1981 400 mg Twice Daily (Bid) | AZD1981 1000 mg Twice Daily (Bid) | Placebo
Started | 95 | 90 | 92 | 91
Completed | 92 | 87 | 86 | 85
Not Completed | 3 | 3 | 6 | 6
Not completed — Adverse Event | 3 | 2 | 5 | 4
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 1
Not completed — Palm stopped to work | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD1981 50 mg Twice Daily (Bid) | AZD1981 400 mg Twice Daily (Bid) | AZD1981 1000 mg Twice Daily (Bid) | Placebo | Total
Number analyzed (Participants) | 95 | 90 | 92 | 91 | 368
Age, Continuous [Mean (Full Range); unit: Years] | 43.3 [18 to 76] | 43 [18 to 79] | 43.5 [18 to 77] | 45.7 [18 to 77] | 44.35 [18 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 19 | 34 | 33 | 113
  Male | 68 | 71 | 58 | 58 | 255

OUTCOME MEASURES:

1. Primary Outcome: Morning Peak Expiratory Flow (mPEF)
Description: Mean mPEF during the treatment period (mean of the last 2 weeks of the treatment period)
Time Frame: Week 4
Population: The efficacy analysis is based on 368 total randomized patients with available data. However, not all patients will have valid, non-missing values for a given outcome measure.
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | AZD1981 50 mg Twice Daily (Bid) | AZD1981 400 mg Twice Daily (Bid) | AZD1981 1000 mg Twice Daily (Bid) | Placebo
Number analyzed (Participants) | 95 | 89 | 92 | 90
L/min | 346.42 (132.70) [-245 to 334] | 362.54 (134.69) [-131 to 213] | 352.87 (124.22) [-158 to 219] | 329.75 (140.14) [-283 to 158]

2. Secondary Outcome: Evening Peak Expiratory Flow (ePEF)
Description: Mean ePEF during the treatment period (mean of the last 2 weeks of the treatment period)
Time Frame: Week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/min
Arm/Group | AZD1981 50 mg Twice Daily (Bid) | AZD1981 400 mg Twice Daily (Bid) | AZD1981 1000 mg Twice Daily (Bid) | Placebo
Number analyzed (Participants) | 95 | 89 | 92 | 91
L/min | 359.83 (129.23) [-192 to 315] | 378.98 (134.54) [-179 to 262] | 368.70 (124.08) [-149 to 225] | 348.87 (142.92) [-202 to 197]

3. Secondary Outcome: Morning Forced Expiratory Volume in 1 Second (mFEV1)
Description: Mean mFEV1 during the treatment period (mean of the last 2 weeks of the treatment period)
Time Frame: Week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L
Arm/Group | AZD1981 50 mg Twice Daily (Bid) | AZD1981 400 mg Twice Daily (Bid) | AZD1981 1000 mg Twice Daily (Bid) | Placebo
Number analyzed (Participants) | 67 | 63 | 71 | 71
L | 2.45 (0.99) [-1.24 to 1.80] | 2.65 (1.03) [-1.41 to 1.04] | 2.53 (0.97) [-0.503 to 0.843] | 2.31 (1.05) [-2.21 to 1.12]

4. Secondary Outcome: Evening Forced Expiratory Volume in 1 Second (eFEV1)
Description: Mean eFEV1 during the treatment period (mean of the last 2 weeks of the treatment period)
Time Frame: Week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L
Arm/Group | AZD1981 50 mg Twice Daily (Bid) | AZD1981 400 mg Twice Daily (Bid) | AZD1981 1000 mg Twice Daily (Bid) | Placebo
Number analyzed (Participants) | 66 | 66 | 73 | 72
L | 2.47 (0.95) [-0.834 to 1.17] | 2.72 (1.02) [-1.56 to 1.20] | 2.63 (0.98) [-0.765 to 2.03] | 2.43 (1.06) [-1.46 to 1.66]

5. Secondary Outcome: Total Use of Reliever
Description: Mean total reliever use during the treatment period (mean of the last 2 weeks of the treatment period)
Time Frame: Week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Number of inhalations per day
Arm/Group | AZD1981 50 mg Twice Daily (Bid) | AZD1981 400 mg Twice Daily (Bid) | AZD1981 1000 mg Twice Daily (Bid) | Placebo
Number analyzed (Participants) | 95 | 90 | 92 | 91
Number of inhalations per day | 2.870 (2.475) [-4.80 to 5.34] | 2.640 (2.303) [-6.36 to 6.59] | 2.569 (2.210) [-8.30 to 3.23] | 2.855 (2.430) [-6.79 to 2.84]

6. Secondary Outcome: Night-time Asthma Symptom Score
Description: Mean night-time asthma symptom score during the treatment period (mean of the last 2 weeks of the treatment period). Scores range from 0 (none) to 3 (bad).
Time Frame: Week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | AZD1981 50 mg Twice Daily (Bid) | AZD1981 400 mg Twice Daily (Bid) | AZD1981 1000 mg Twice Daily (Bid) | Placebo
Number analyzed (Participants) | 95 | 90 | 92 | 91
Scores on a scale | 0.998 (0.633) [-2.80 to 0.733] | 0.881 (0.543) [-1.36 to 0.786] | 0.912 (0.594) [-1.83 to 0.655] | 1.008 (0.614) [-2.12 to 0.714]

7. Secondary Outcome: Day-time Asthma Symptom Score
Description: Mean day-time asthma symptom score during the treatment period (mean of the last 2 weeks of the treatment period). Scores range from 0 (none) to 3 (bad).
Time Frame: Week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | AZD1981 50 mg Twice Daily (Bid) | AZD1981 400 mg Twice Daily (Bid) | AZD1981 1000 mg Twice Daily (Bid) | Placebo
Number analyzed (Participants) | 95 | 90 | 92 | 91
Scores on a scale | 1.037 (0.609) [-2.80 to 0.850] | 0.933 (0.556) [-1.00 to 1.04] | 0.995 (0.552) [-2.20 to 1.25] | 1.105 (0.645) [-2.00 to 1.62]

8. Secondary Outcome: Awakenings
Description: Mean percentage of awakenings due to asthma symptoms during the treatment period (mean of the last 2 weeks of the treatment period)
Time Frame: Week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of days
Arm/Group | AZD1981 50 mg Twice Daily (Bid) | AZD1981 400 mg Twice Daily (Bid) | AZD1981 1000 mg Twice Daily (Bid) | Placebo
Number analyzed (Participants) | 95 | 90 | 92 | 91
Percentage of days | 38.59 (40.25) [-100 to 44.4] | 33.18 (38.93) [-84.6 to 100] | 33.34 (37.68) [-92.3 to 60] | 37.32 (39.51) [-100 to 58.6]

9. Secondary Outcome: Asthma Control Day
Description: Mean percentage of asthma control days during the treatment period (mean of the last 2 weeks of the treatment period). An asthma control day is defined as a symptom-free day with no use of reliever medication during day and night. A symptom-free day is defined as a day and a night with no asthma symptoms and a day and night with no awakenings due to asthma symptoms.
Time Frame: Week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of days
Arm/Group | AZD1981 50 mg Twice Daily (Bid) | AZD1981 400 mg Twice Daily (Bid) | AZD1981 1000 mg Twice Daily (Bid) | Placebo
Number analyzed (Participants) | 95 | 90 | 92 | 91
Percentage of days | 10.78 (25.79) [-12.5 to 100] | 7.48 (20.71) [-20 to 100] | 13.23 (26.24) [-38.3 to 100] | 10.08 (22.36) [-1.67 to 100]

10. Secondary Outcome: Symptom Free Day
Description: Mean percentage of symptom free days during the treatment period (mean of the last 2 weeks of the treatment period). A symptom-free day is defined as a day and a night with no asthma symptoms and a day and night with no awakenings due to asthma symptoms.
Time Frame: Week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of days
Arm/Group | AZD1981 50 mg Twice Daily (Bid) | AZD1981 400 mg Twice Daily (Bid) | AZD1981 1000 mg Twice Daily (Bid) | Placebo
Number analyzed (Participants) | 95 | 90 | 92 | 91
Percentage of days | 17.33 (32.16) [-49.2 to 100] | 13.95 (28.35) [-52.3 to 100] | 15.56 (28.51) [-72.3 to 100] | 14.31 (26.28) [-23.8 to 100]

11. Secondary Outcome: Reliever Free Day
Description: Mean percentage of reliever free days during the treatment period (mean of the last 2 weeks of the treatment period). A reliever free day is defined as a day and a night with no use of as-needed medication.
Time Frame: Week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percentage of days
Arm/Group | AZD1981 50 mg Twice Daily (Bid) | AZD1981 400 mg Twice Daily (Bid) | AZD1981 1000 mg Twice Daily (Bid) | Placebo
Number analyzed (Participants) | 95 | 90 | 92 | 91
Percentage of days | 22.59 (34.57) [-16.9 to 100] | 20.60 (32.01) [-30.0 to 100] | 24.13 (32.12) [-50.0 to 100] | 20.94 (32.97) [-23.6 to 100]

12. Secondary Outcome: Forced Expiratory Volume in 1 Second (FEV1) at the Clinic
Description: Mean FEV1 during the treatment period (mean value at Week 4)
Time Frame: Week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L
Arm/Group | AZD1981 50 mg Twice Daily (Bid) | AZD1981 400 mg Twice Daily (Bid) | AZD1981 1000 mg Twice Daily (Bid) | Placebo
Number analyzed (Participants) | 93 | 90 | 92 | 88
L | 2.653 (1.051) [-0.760 to 2.02] | 2.739 (1.028) [-0.730 to 2.16] | 2.628 (1.057) [-2.46 to 2.04] | 2.400 (0.945) [-0.740 to 1.26]

13. Secondary Outcome: Forced Vital Capacity (FVC) at the Clinic
Description: Mean FVC during the treatment period (mean value at Week 4)
Time Frame: Week 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L
Arm/Group | AZD1981 50 mg Twice Daily (Bid) | AZD1981 400 mg Twice Daily (Bid) | AZD1981 1000 mg Twice Daily (Bid) | Placebo
Number analyzed (Participants) | 93 | 90 | 92 | 88
L | 3.704 (1.268) [-1.48 to 2.21] | 3.892 (1.295) [-0.980 to 2.30] | 3.546 (1.257) [-1.03 to 2.68] | 3.563 (1.215) [-0.990 to 2.02]

14. Secondary Outcome: Asthma Control Questionnaire 5 Items (ACQ5)
Description: Mean ACQ5 score during the treatment period (mean value at Week 4). Scores range from 0 (good) to 6 (poor control).
Time Frame: Week 4
Population: as for outcome 1
Measure: Mean (Full Range); unit: Scores on a scale
Arm/Group | AZD1981 50 mg Twice Daily (Bid) | AZD1981 400 mg Twice Daily (Bid) | AZD1981 1000 mg Twice Daily (Bid) | Placebo
Number analyzed (Participants) | 92 | 89 | 86 | 85
Scores on a scale | 1.69 (-2.40) [0 to 4.00] | 1.58 (-2.40) [0 to 3.80] | 1.64 (-3.20) [0 to 4.60] | 1.91 (-2.60) [0 to 4.20]

15. Secondary Outcome: Adverse Event (AE)
Description: Number of patients reporting at least one event
Time Frame: 4 weeks
Measure: Number; unit: Participants
Arm/Group | AZD1981 50 mg Twice Daily (Bid) | AZD1981 400 mg Twice Daily (Bid) | AZD1981 1000 mg Twice Daily (Bid) | Placebo
Number analyzed (Participants) | 95 | 90 | 92 | 91
Participants | 28 | 22 | 33 | 24

ADVERSE EVENTS:
Arm/Group | AZD1981 50 mg Twice Daily (Bid) | AZD1981 400 mg Twice Daily (Bid) | AZD1981 1000 mg Twice Daily (Bid) | Placebo
Serious Adverse Events (participants affected / at risk) | 0/95 | 0/90 | 1/92 | 1/91
Other Adverse Events (participants affected / at risk) | 5/95 | 6/90 | 11/92 | 7/91
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AZD1981 50 mg Twice Daily (Bid) (N=95) | AZD1981 400 mg Twice Daily (Bid) (N=90) | AZD1981 1000 mg Twice Daily (Bid) (N=92) | Placebo (N=91)
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AZD1981 50 mg Twice Daily (Bid) (N=95) | AZD1981 400 mg Twice Daily (Bid) (N=90) | AZD1981 1000 mg Twice Daily (Bid) (N=92) | Placebo (N=91)
Gastritis (Gastrointestinal disorders) | 1 | 2 | 5 | 3
Headache (Nervous system disorders) | 2 | 4 | 3 | 2
Asthma (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 3 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less